CLINICAL TRIAL: NCT00984815
Title: Open-Label Safety Study of HZT-501 in Patients Who Require Long-Term Daily Non-Steroidal Anti-Inflammatory Drug Treatment
Brief Title: Safety Study of HZT-501 in Patients Who Require Long-Term Daily Non-steroidal Anti-inflammatory Drug Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZ-CA-401
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Results first posted 2013-07-25 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Chronic Low Back Pain; Chronic Regional Pain Syndrome; Chronic Soft Tissue Pain
Keywords: NSAID; Chronic Pain; Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Complex Regional Pain Syndromes; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HZT-501 (Experimental): Open-label treatment with HZT-501
  Interventions: Drug: HZT-501

INTERVENTIONS:
Drug: HZT-501 — Fixed-dose combination oral tablet 800mg Ibuprofen/26.6 mg Famotidine taken three times per day

SUMMARY:
The purpose of this study is to evaluate the safety of long-term treatment with HZT-501, a fixed-dose combination oral tablet of 800 mg ibuprofen and 26.6 mg famotidine for patients that require long-term NSAID treatment.

DETAILED DESCRIPTION:
HZT-501, a fixed-dose combination of ibuprofen, a pain and inflammation relieving non-steroidal anti-inflammatory drug (NSAID), and famotidine, a histamine type 2 receptor antagonist (H2RA), is being developed for the treatment of patients with signs and symptoms of osteoarthritis, rheumatoid arthritis, mild to moderate pain or dysmenorrhea who are at risk of developing ibuprofen-associated upper gastrointestinal ulcers.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Patient is capable of understanding the purpose and risks of the study and is able to provide written Informed Consent.
* Patient is male or female, aged 40 to 80 years of age.
* Patient is expected to require daily administration of an NSAID for at least the coming year for conditions including but not limited to: osteoarthritis, rheumatoid arthritis, chronic low back pain, chronic regional pain syndrome, chronic soft tissue pain.
* Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use medically acceptable methods of contraception throughout the entire study period.
* Patient is willing and able to comply with the prescribed treatment protocol and evaluations.

Exclusion Criteria:

* Patient has a history of or experienced any of the following:
* NSAID-associated and/or primary peptic ulcer disease-associated serious gastrointestinal complications such as perforation of ulcers, gastric outlet obstruction due to ulcers, and/or acute gastrointestinal bleeding
* NSAID-induced asthma exacerbation, acute renal failure, interstitial nephritis, and/or hepatitis
* Malignant disease of the gastrointestinal tract
* Erosive esophagitis
* Coronary artery bypass graft (CABG) surgery within the 14 days prior to study Day 0
* Uncontrolled diabetes mellitus as evidenced by Hemoglobin A1c > 7%
* Known history of human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C
* Patient has active cardiac, renal, and/or hepatic disease, as evidenced by:
* Creatinine clearance < 45 mL/min (based on the Cockroft-Gault formula) at Screening
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal at Screening
* History of acute myocardial infarction, unstable cardiac arrhythmias, and/or stroke within the 6 months prior to study entry
* Uncontrolled congestive heart failure
* Uncontrolled hypertension
* Patient currently is participating in an investigational drug study, or patient participated in an investigational drug study within the 30 days prior to study entry.
* Female patient has a positive urine pregnancy test at Screening and/or Study Day 0.
* Patient has a concomitant disease or condition that, in the opinion of the Investigator, could interfere with the conduct of the study or could put the patient at unacceptable risk.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - University of Illinois Medical Center, Department of Medicine, Chicago, Illinois
  - Illinois Bone & Joint Institute, Morton Grove, Illinois
  - Altoona Center for Clinical Research Altoona Arthritis, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas

REFERENCES:
- [Derived] Bello AE, Kent JD, Grahn AY, Ball J, Holt RJ. One-year open-label safety evaluation of the fixed combination of ibuprofen and famotidine with a prospective analysis of dyspepsia. Curr Med Res Opin. 2015 Mar;31(3):397-405. doi: 10.1185/03007995.2014.999152. Epub 2015 Jan 9. PMID 25495134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 100 eligible participants were to be enrolled at 4 U.S. study centers (3 private practice rheumatology centers and 1 academic center) between September, 2009 and June, 2010.
Pre-assignment Details: Eligible participants, 40-80 years of age inclusive, expected to require daily administration of a non-steroidal anti-inflammatory drug (NSAID) for at least the coming 12 months were enrolled. Of the approximately 100 participants enrolled, it was expected that at least 30 would complete the 54-week treatment period.
Groups:
- HZT-501: Open-label treatment with HZT-501(ibuprofen 800 mg/famotidine 26.6 mg) tablets. All doses of study drug will be self-administered orally 3 times daily (TID), for up to 54 weeks.
Period: Overall Study
Arm/Group | HZT-501
Started | 86
Completed | 56
Not Completed | 30

BASELINE CHARACTERISTICS:
Groups:
- HZT-501: Open-label treatment with HZT-501 (ibuprofen 800 mg/famotidine 26.6 mg) tablets self-administered orally three times daily (TID) for up to 54 weeks.
Arm/Group | HZT-501
Number analyzed (Participants) | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 69
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 86

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in the Pain Intensity Scale of the Severity of Dyspepsia Assessment (SODA) Questionnaire at 54 Weeks
Description: The pain intensity scale of the SODA questionnaire ranges from 2 - 47. Change from baseline compares the score at Week 54 to the baseline score for each participant who completed the pain intensity questions of the SODA questionnaire at baseline and Week 54. Higher scores indicate greater symptom severity and therefore a negative mean change from baseline is indicative of an improvement in symptoms.
Time Frame: Baseline and 54 Weeks
Population: 54 participants who completed the pain intensity questions of the SODA questionnaire at baseline and Week 54.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | HZT-501
Number analyzed (Participants) | 54
Scores on a scale | -3.22 (10.522)

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Time Frame: 54 weeks
Population: All participants enrolled and who received at least one dose of study drug comprised the Safety Population.
Measure: Number; unit: participants
Arm/Group | HZT-501
Number analyzed (Participants) | 86
participants | 76

3. Secondary Outcome: Change From Baseline in the Non-pain Symptoms Scale of the Severity of Dyspepsia Assessment (SODA) Questionnaire at 54 Weeks
Description: The non-pain symptom scale of the SODA questionnaire ranges from 7 - 35. Change from baseline compares the score at Week 54 to the baseline score for each participant that completed the non-pain symptom questions of the SODA questionnaire at baseline and Week 54. Higher scores indicate greater symptom severity and therefore a negative mean change from baseline is indicative of an improvement in symptoms.
Time Frame: Baseline and 54 Weeks
Population: 55 participants who completed the non-pain symptom questions of the SODA questionnaire at baseline and Week 54.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | HZT-501
Number analyzed (Participants) | 55
Scores on a scale | -1.44 (3.934)

4. Secondary Outcome: Change From Baseline in the Satisfaction With Dyspepsia-Related Health Scale of the Severity of Dyspepsia Assessment (SODA) Questionnaire at 54 Weeks
Description: The satisfaction with dyspepsia-related health scale of the SODA questionnaire ranges from 2 - 23. Change from baseline compares the score at Week 54 to the baseline score for each participant who completed the Satisfaction questions of the SODA questionnaire at baseline and Week 54. A positive change from baseline in the SODA satisfaction scale represents a participant's overall improved satisfaction with their dyspepsia-related health.
Time Frame: Baseline and 54 Weeks
Population: 55 participants who completed the satisfaction with dyspepsia-related health questions of the SODA questionnaire at baseline and week 54.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | HZT-501
Number analyzed (Participants) | 55
Scores on a scale | 2.69 (5.504)

ADVERSE EVENTS:
Arm/Group | HZT-501
Serious Adverse Events (participants affected / at risk) | 9/86
Other Adverse Events (participants affected / at risk) | 76/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HZT-501 (N=86)
angina unstable (Cardiac disorders) | 1
gastric ulcer (Gastrointestinal disorders) | 1
small intestinal obstruction (Gastrointestinal disorders) | 1
cellulitis staphylococcal (Infections and infestations) | 1
escherichia sepsis (Infections and infestations) | 1
pyelonephritis (Infections and infestations) | 1
back pain (Musculoskeletal and connective tissue disorders) | 1
convulsion (Nervous system disorders) | 1
global amnesia (Nervous system disorders) | 1
depression (Psychiatric disorders) | 1
renal failure acute (Renal and urinary disorders) | 1
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HZT-501 (N=86)
abdominal distension (Gastrointestinal disorders) | 10
dyspepsia (Gastrointestinal disorders) | 10
flatulence (Gastrointestinal disorders) | 9
diarrhoea (Gastrointestinal disorders) | 8
nausea (Gastrointestinal disorders) | 8
abdominal pain lower (Gastrointestinal disorders) | 4
constipation (Gastrointestinal disorders) | 4
gastroesophageal reflux disease (Gastrointestinal disorders) | 4
abdominal pain (Gastrointestinal disorders) | 3
abdominal pain upper (Gastrointestinal disorders) | 3
vomiting (Gastrointestinal disorders) | 3
oedema peripheral (Gastrointestinal disorders) | 4
pitting oedema (General disorders) | 3
sinusitis (Infections and infestations) | 9
urinary tract infection (Infections and infestations) | 8
gastroenteritis viral (Infections and infestations) | 7
upper respiratory tract infection (Infections and infestations) | 7
influenza (Infections and infestations) | 4
herpes zoster (Infections and infestations) | 3
excoriation (Injury, poisoning and procedural complications) | 5
muscle strain (Injury, poisoning and procedural complications) | 4
procedural pain (Injury, poisoning and procedural complications) | 4
arthralgia (Musculoskeletal and connective tissue disorders) | 5
back pain (Musculoskeletal and connective tissue disorders) | 4
osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
headache (Nervous system disorders) | 3
depression (Psychiatric disorders) | 3
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4
dermatitis contact (Skin and subcutaneous tissue disorders) | 3
rash (Skin and subcutaneous tissue disorders) | 3
hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may disclose data resulting from the study upon the earliest of: a) publication of a multi-center publication coordinated by Sponsor, b) submission of the data by Sponsor to the FDA, and c) 18 months after the study is completed at all sites if a multi-center publication is not submitted by Sponsor for publication provided PI submits proposed publication at least 60 days in advance for review of any Sponsor Confidential Information.